CLINICAL TRIAL: NCT01810016
Title: Phase I Study of NY-ESO-1 Vaccine in Combination With Ipilimumab in Patients With Unresectable or Metastatic Melanoma, for Whom Treatment With Ipilimumab is Indicated
Brief Title: NY-ESO-1 Vaccine in Combination With Ipilimumab in Patients With Unresectable or Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment due to change in standard of care
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Cancer Research Institute, NY, USA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2012-004
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Unresectable or Metastatic Melanoma
Keywords: NY-ESO-1; Metastatic Melanoma; Ipilimumab; Phase I; Adjuvant; Immunologic; Vaccination; Immunotherapy; Neoplasm
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Ipilimumab; poly ICLC; Monatide (IMS 3015)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Ipilimumab (IV) followed by NY-ESO-1 recombinant protein mixed with Poly-ICLC and Montanide (SC) every 3 weeks for 4 doses.
  Interventions: Biological: Ipilimumab; Biological: NY-ESO-1 Protein Vaccine
- Arm B (Experimental): Ipilimumab (IV) followed by NY-ESO-1 OLP4 mixed with Poly-ICLC and Montanide (SC) every 3 weeks for 4 doses.
  Interventions: Biological: Ipilimumab; Biological: NY-ESO-1 OLP4 Vaccine with Poly-ICLC and Montanide
- Arm C (Experimental): Ipilimumab (IV) followed by NY-ESO-1 OLP4 mixed with Poly-ICLC (SC) every 3 weeks for 4 doses.
  Interventions: Biological: Ipilimumab; Biological: NY-ESO-1 OLP4 Vaccine with Poly-ICLC

INTERVENTIONS:
Biological: Ipilimumab — Ipilimumab was administered IV over 90 minutes at a dose of 3 mg/kg directly preceding the NY-ESO-1 injection every 3 weeks for 4 doses.
  Other Names: Yervoy
Biological: NY-ESO-1 Protein Vaccine — NY-ESO-1 recombinant protein (250 µg) was mixed with Poly-ICLC (1 mg) and Montanide ISA-51 VG (1 mL) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
  Arms: Arm A
Biological: NY-ESO-1 OLP4 Vaccine with Poly-ICLC and Montanide — NY-ESO-1 OLP4 (1 mg) was mixed in 5% dextrose solution in water with Poly-ICLC (1 mg) and Montanide ISA-51 VG (1 mL) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
  Arms: Arm B
Biological: NY-ESO-1 OLP4 Vaccine with Poly-ICLC — NY-ESO-1 OLP4 (1 mg) was mixed in 5% dextrose solution in water with Poly-ICLC (1 mg) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
  Arms: Arm C

SUMMARY:
This was a Phase 1, open-label, non-randomized study of the combination of NY-ESO-1 plus ipilimumab in patients with unresectable or metastatic melanoma for whom treatment with ipilimumab was indicated. Patients must have had evidence of NY-ESO-1 or LAGE-1 tumor positivity and radiologically measurable disease by the immune-related Response Criteria (irRC). Primary study objectives were to determine the safety and tolerability of the combination and to evaluate humoral and cellular immune response. Secondary objectives were to evaluate tumor response and immunological changes in the tumor microenvironment.

DETAILED DESCRIPTION:
Patients were enrolled sequentially, alternating among 3 treatment arms. Study treatment comprised ipilimumab 3 mg/kg administered intravenously (IV) over 90 minutes every 3 weeks for 4 doses followed by the NY-ESO-1 vaccine administered subcutaneously (SC). Arm A received the NY-ESO-1 recombinant protein mixed with polyinosinic-polycytidylic acid-poly-L-lysine carboxymethylcellulose (Poly-ICLC) and Montanide; Arm B received NY-ESO-1 overlapping long peptides 4 (OLP4) mixed with Poly-ICLC and Montanide; and Arm C received NY-ESO-1 OLP4 mixed with Poly-ICLC (without Montanide). The vaccine was administered immediately following the ipilimumab infusion, and patients were observed for 1 hour following administration. No dose adjustments or delays were permitted.

Because the study treatment regimens had not been previously investigated in humans, the first patient in each treatment arm was followed for 28 days and evaluated for any regimen-limiting toxicity (RLT), defined as any dose-limiting toxicity (DLT) that could not be attributed solely to either the vaccine or ipilimumab and was therefore considered to be related to the combination. If an RLT was observed in the first patient, the second patient was to be evaluated for 28 days before the third patient was enrolled. If at any point ≥ 2 RLTs were observed in a treatment arm, accrual to that arm was to be terminated and the combination in that arm was to be declared unsafe.

Patients were monitored for safety, immune and tumor response, and immunological changes in the tumor microenvironment for the duration of study participation, which may have been up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable or metastatic melanoma, for whom treatment with ipilimumab was indicated as per ipilimumab/Yervoy® package insert (applicable for United States [US] sites) or product information (applicable for Australia site).
2. Radiologically measurable disease by irRC.
3. Tumor expression of NY-ESO-1 or LAGE-1 antigen by immunohistochemistry or reverse transcriptase-polymerase chain reaction (RT-PCR), or evidence of seropositivity to NY-ESO-1 or LAGE-1.
4. Willingness to provide at least one pre-and post-vaccination tumor biopsy sample.
5. Expected survival of at least 4 months.
6. At the time of Day 1 of the study, patients must have been at least 3 weeks since surgery.
7. At the time of Day 1 of the study, patients with brain metastases must have been asymptomatic and:

   * at least 8 weeks without tumor progression after any whole brain radiotherapy;
   * at least 4 weeks since craniotomy and resection or stereotactic radiosurgery;
   * at least 3 weeks without new brain metastases as evidenced by magnetic resonance imaging (MRI).
8. Eastern Cooperative Oncology Group performance status of 0 to 2.
9. Laboratory parameters for vital functions must have been in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which must have been within the ranges specified:

   * hemoglobin: ≥ 10 g/dL;
   * neutrophil count: ≥ 1.5 x 10^9/L;
   * lymphocyte count: ≥ lower limit of normal (LLN);
   * platelet count: ≥ 80 x 10^9/L;
   * serum creatinine: ≤ 2 mg/dL;
   * serum bilirubin: ≤ 2 x upper limit of normal (ULN);
   * aspartate aminotransferase (AST)/alanine aminotransferase (ALT): ≤ 2 x ULN.
10. Had been informed of other treatment options.
11. Age ≥ 18 years.
12. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Any contraindications for ipilimumab/Yervoy® as per package insert (applicable for US sites) or product information (applicable for Australia site).
2. Prior exposure to NY-ESO-1 vaccine.
3. Active autoimmune disease, symptoms or conditions except for vitiligo, type I diabetes, treated thyroiditis, asymptomatic laboratory evidence of autoimmune disease (e.g., +antinuclear antibody [ANA], +rheumatoid factor [RF], antithyroglobulin antibodies), or mild arthritis requiring no therapy or manageable with nonsteroidal anti-inflammatory drugs (NSAIDs).
4. Unresolved immune-related adverse events following prior biological therapy.
5. Systemic treatment with high-dose corticosteroids (greater than prednisone 10 mg daily or equivalent).
6. Treatment with protocol-specified non-permitted concomitant therapies.
7. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may have been available.
8. Myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, chest pain or shortness of breath with activity, or other heart conditions being treated by a doctor.
9. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
10. Known immunodeficiency or human immunodeficiency virus positivity, active Hepatitis B or active Hepatitis C.
11. History of severe allergic reactions to vaccines or unknown allergens.
12. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
13. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to Day 1 of the study.
14. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
15. Lack of availability for immunological and clinical follow-up assessments.
16. Women who were breast feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) done within 14 days prior to first dosing and urine test within 72 hours prior to first dosing.
17. Women of childbearing potential not using a medically acceptable means of contraception for the duration of the study.
18. Any condition that, in the clinical judgment of the treating physician, was likely to prevent the patient from complying with any aspect of the protocol or that may have put the patient at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Postow, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Hassane M Zarour, MD, Principal Investigator — University of Pittsburgh; Craig L Slingluff, MD, Principal Investigator — University of Virginia; Jonathan Cebon, MBBS, FRACP, PhD, Principal Investigator — Austin Health, Ludwig Oncology Unit; Philip Friedlander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (4):
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Center, Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
- Austin Health, Ludwig Oncology Unit, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Ipi, NY-ESO-1 Protein): Ipilimumab was administered IV over 90 minutes at a dose of 3 mg/kg directly preceding the NY-ESO-1 injection every 3 weeks for 4 doses.
  NY-ESO-1 recombinant protein (250 µg) was mixed with Poly-ICLC (1 mg) and Montanide ISA-51 VG (1 mL) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
- Arm B (Ipi, NY-ESO-1 OLP4): Ipilimumab was administered IV over 90 minutes at a dose of 3 mg/kg directly preceding the NY-ESO-1 injection every 3 weeks for 4 doses.
  NY-ESO-1 OLP4 (1 mg) was mixed in 5% dextrose solution in water with Poly-ICLC (1 mg) and Montanide ISA-51 VG (1 mL) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
- Arm C (Ipi, NY-ESO-1 OLP4): Ipilimumab was administered IV over 90 minutes at a dose of 3 mg/kg directly preceding the NY-ESO-1 injection every 3 weeks for 4 doses.
  NY-ESO-1 OLP4 (1 mg) was mixed in 5% dextrose solution in water with Poly-ICLC (1 mg) and administered SC directly following the ipilimumab infusion every 3 weeks for 4 doses.
Period: Overall Study
Arm/Group | Arm A (Ipi, NY-ESO-1 Protein) | Arm B (Ipi, NY-ESO-1 OLP4) | Arm C (Ipi, NY-ESO-1 OLP4)
Started | 5 | 2 | 1
Completed | 4 | 1 | 0
Not Completed | 1 | 1 | 1
Not completed — Progressive disease | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ipi, NY-ESO-1 Protein) | Arm B (Ipi, NY-ESO-1 OLP4) | Arm C (Ipi, NY-ESO-1 OLP4) | Total
Number analyzed (Participants) | 5 | 2 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.7) | 61.5 (7.8) | 71.0 (NA) — Only 1 patient is included in this arm so a standard deviation is not calculable. | 63.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 4 | 2 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 2 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 1 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI was not available for 1 patient in Arm A.
  kg/m^2
    number analyzed (Participants) | 4 | 2 | 1 | 7
    (all) | 36.6 (11.5) | 26.2 (0.2) | 29.0 (NA) — Only 1 patient is included in this arm so a standard deviation is not calculable. | 32.5 (9.6)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — grade 0: fully active, able to carry on pre-disease performance without restriction.
  grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work.
  grade 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours.
  grade 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  grade 4: completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  grade 5: dead.
  Participants
    0 | 3 | 1 | 0 | 4
    1 | 2 | 1 | 1 | 4
Tumor Stage at Study Entry [Count of Participants; unit: Participants] — The American Joint Committee on Cancer staging system is used to stage melanoma based on the Tumor, Node, Metastasis (TNM) system. The melanoma tumor stage represents a composite score that accounts for the thickness and ulceration of the primary tumor (T), presence and extent of metastasis to regional lymph nodes (N), and presence and extent of distant metastases (M). Stage IIIC indicates advanced melanoma that has metastasized to the regional lymph nodes, and Stage IV indicates metastasis to distant lymph nodes and/or other organs/tissue.
  Participants
    IIIC | 1 | 0 | 0 | 1
    IV | 4 | 2 | 1 | 7
Antigen [Count of Participants; unit: Participants]
  NY-ESO-1 | 1 | 2 | 0 | 3
  LAGE-1 | 0 | 0 | 0 | 0
  None | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period. Dose-limiting toxicity (DLT) was defined as any ≥ Grade 3 hematologic or non-hematologic toxicity that was definitely, probably, or possibly related to the administration of the NY-ESO-1 vaccine or as any toxicity that was definitely, probably, or possibly related to ipilimumab and required permanent discontinuation of ipilimumab in accordance with local prescribing information. DLT assessments were based on the combination of all vaccine components, not on the components individually.
Time Frame: Continuously for up to 6 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipi, NY-ESO-1 Protein) | Arm B (Ipi, NY-ESO-1 OLP4) | Arm C (Ipi, NY-ESO-1 OLP4)
Number analyzed (Participants) | 5 | 2 | 1
Participants
  Any TEAE | 5 | 2 | 1
  Maximum grade 1 TEAE | 1 | 1 | 0
  Maximum grade 2 TEAE | 2 | 1 | 0
  Maximum grade 3 TEAE | 2 | 0 | 0
  Maximum grade 4 TEAE | 0 | 0 | 0
  Maximum grade 5 TEAE | 0 | 0 | 1
  NY-ESO-1-related TEAE | 4 | 2 | 0
  Ipilimumab-related TEAE | 5 | 2 | 0
  Serious TEAE | 2 | 0 | 1
  TEAE Leading to Treatment Discontinuation | 0 | 0 | 1
  TEAE Meeting DLT Criteria | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Immune-related Tumor Response at the Last Assessment
Description: Immune-related tumor response was evaluated using the imaging techniques considered appropriate by the Investigators at Baseline, Week 13, and at the end of the study (Week 20 ± 1 week). Tumor response was designated according to the immune-related Response Criteria (irRC) (Wolchok et al. Clin Cancer Res 2009;15:7412-20) into the following categories: immune-related complete response (irCR) requires disappearance of all lesions in two consecutive observations not less than 4 weeks apart; immune-related partial response (irPR) requires ≥ 50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart; immune-related stable disease (irSD) is assigned when neither a 50% decrease from baseline tumor burden nor a 25% increase in tumor burden from nadir can be established; immune-related progressive disease (irPD) requires a ≥ 25% increase from nadir in tumor burden at any single time point in two consecutive observations at least 4 weeks apart.
Time Frame: Up to 5 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipi, NY-ESO-1 Protein) | Arm B (Ipi, NY-ESO-1 OLP4) | Arm C (Ipi, NY-ESO-1 OLP4)
Number analyzed (Participants) | 5 | 2 | 1
Participants
  irSD at Last Assessment | 4 | 0 | 0
  irPD at Last Assessment | 0 | 2 | 0
  Not evaluated | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 6 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.0), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | Arm A (Ipi, NY-ESO-1 Protein) | Arm B (Ipi, NY-ESO-1 OLP4) | Arm C (Ipi, NY-ESO-1 OLP4)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipi, NY-ESO-1 Protein) (N=5) | Arm B (Ipi, NY-ESO-1 OLP4) (N=2) | Arm C (Ipi, NY-ESO-1 OLP4) (N=1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipi, NY-ESO-1 Protein) (N=5) | Arm B (Ipi, NY-ESO-1 OLP4) (N=2) | Arm C (Ipi, NY-ESO-1 OLP4) (N=1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 1
Injection site reaction (General disorders) | 4 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Chills (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Xerosis (General disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Scleral discolouration (Eye disorders) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
As the study was terminated early due to slow enrollment, immune response (humoral and cellular) analyses were not performed as outlined in the protocol due to small sample sizes within each arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less